CLINICAL TRIAL: NCT06368999
Title: Neurophysiological and Neuropsychological Evalution in Healthcare Workers of Stress Condition
Brief Title: Neurophysiological and Neuropsychological Evalution in Healthcare Workers
Acronym: EEGCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EEGCOV
Record Dates: First submitted 2024-03-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: study of brain EEG activity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- heatlhcare workers (Experimental)
  Interventions: Diagnostic Test: EEG

INTERVENTIONS:
Diagnostic Test: EEG — registration of 8 minutes of EEG

SUMMARY:
The goal of this observational study is to compare in participant population the effect of stress condition on cerebral EEG activity Participants will do an 8 minutes EEG registration. Researchers will compare EEG activity of heathcare workers.

ELIGIBILITY:
Inclusion Criteria:

* healthcare workers

Exclusion Criteria:

* neurological disorders

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
EEG activity | immediately after the outbreak of the pandemic (first session) and almost 6 months later (second session).
  The subjects were instrumented with 19 bridge silver and silver chloride electrodes fitted on a plastic prewired head cap and placed on the scalp according to the 10-20 system (namely: Fp1, Fp2, F3, F4, F7, F8, Fz, C3, C4, Cz, P3, P4, Pz, T3, T4, T5, T6, O1, and O2), with an electroconductive paste applied between the electrodes and the skin to guarantee optimal connection The signals were recorded with a 512 Hz sampling frequency and filtered by an offline first order zero-phase Butterworth band-pass filter, with cutoff frequencies set, respectively, at 1.6 and 70 Hz to remove frequencies outside the range of interest. After this pre-processing, the main EEG rhythms and dominant frequencies were extracted by spectral and connectivity analyses. Delta (1.6-4 Hz), theta (4-8 Hz), alpha (8-13 Hz), beta (13-30 Hz), gamma1 (30-50 Hz), and gamma2 (50-70 Hz) frequency bands were considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No